CLINICAL TRIAL: NCT04838873
Title: Randomised Controlled Trial of Open Versus Laparoscopic Radical Cystectomy at a Laparoscopic Naive Center
Brief Title: Trial of Open Versus Laparoscopic Radical Cystectomy at a Laparoscopic Naive Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelbary Ali, Lecturer of Surgical Oncology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SO1901-31004
Record Dates: First submitted 2021-03-30; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Bladder Cancer; Laparoscopy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Radical Cystectomy (Active Comparator): Standard open radical cystectomy.
  Interventions: Procedure: Open radical cystectomy
- Laparoscopic-assisted radical cystectomy. (Experimental): Laparoscopic-assisted radical cystectomy.
  Interventions: Procedure: Laparoscopic-assisted radical cystectomy

INTERVENTIONS:
Procedure: Open radical cystectomy — Standard open radical cystectomy and urinary diversion
  Arms: Open Radical Cystectomy
Procedure: Laparoscopic-assisted radical cystectomy — Laparoscopic-assisted radical cystectomy and extracorporeal urinary diversion
  Arms: Laparoscopic-assisted radical cystectomy.

SUMMARY:
This study is a prospective randomised controlled study of urinary bladder cancer patients presented to urology unit at National Cancer Institute; Cairo University.

DETAILED DESCRIPTION:
The study will randomise 60 patients to one of two arms; laparoscopic-assisted radical cystectomy and open radical cystectomy. The focus of the study will be a comparison of both approaches on the patients' peri-operative outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with transitional cell carcinoma, squamous cell carcinoma and urinary bladder adenocarcinoma.
* Patients fit for surgery (ECOG Performance Status 0,1).

Exclusion Criteria:

* Patients with medical comorbidities that preclude surgical management or minimally invasive techniques.
* Patients with advanced hydronephrosis or renal failure.
* Patients refusing surgery.
* Patients with urinary bladder cancer invading bladder neck or prostatic urethra.
* Patients with metastatic urinary bladder cancer.
* Patients who received prior pelvic radiotherapy.
* Patients refusing randomization and/or participation in the trial.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Operative time | During surgery
  OR time as measured in minutes, divided into time required to perform the cystectomy, lymph node dissection, and urinary diversion.
Blood loss | During surgery
  EBL as measured in millilitres, including the effluent from the suction canister as well as estimates of the gauze swabs.
Length of hospital stay | Immediate post-operative period.
  LOS as measured in days
Time to oral intake | Immediate post-operative period
  Measured in days
Conversion rate | During surgery
  Rate of conversion from laparoscopy to open surgery
Re-admission rate. | Intra-operative to sixth months.
  Re-hospitalization requirement.
Opioid requirements. | During surgery through first post-operative week.
  Requirement, dose and duration of narcotic analgesia.
Visceral injury | During surgery
  Any organ injury encountered during the operation.
Urine leak | Up to 4 weeks
  Leakage of urine from urinary enteric anastomosis
Wound dehiscence, infection. | Up to 4 weeks
  Wound gaping, evisceration or infection.
Enteric fistula | Up to 4 weeks
  Leakage of intestinal contents due to failure of entero-enteric anastomosis
Sepsis | Up to 4 weeks
  Infection triggering a systematic immune response
Venous thromboembolism | Up to 2 months
  DVT or pulmonary embolism

SECONDARY OUTCOMES:
pT stage | Within 10 days post surgery.
  Pathologic tumor stage (Stage 1, stage 2, stage 3 or stage 4)
Lymph node retrieval | Within 10 days post surgery.
  Number of lymph nodes retrieved by open versus laparoscopic approaches.
pN stage | Within 10 days post surgery.
  Lymph node metastasis (positive or negative), and number of positive nodes if present.
Surgical margins | Within 10 days post surgery
  Positive margins or negative margins. Location of positive margins (Urethral, ureteric)
Histological grade | Within 10 days post surgery
  Low grade, intermediate grade or high grade

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Aboulkassem, M.D., Ph.D., Principal Investigator — National Cancer Institute, Cairo University
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No